CLINICAL TRIAL: NCT06072131
Title: A Phase 3, Randomized, Open-Label Study Comparing the Efficacy and Safety of the Combination of Beleodaq-CHOP or Folotyn-COP to the CHOP Regimen Alone in Newly Diagnosed Patients With Peripheral T-Cell Lymphoma
Brief Title: To Evaluate Efficacy of Belinostat or Pralatrexate in Combination Against CHOP Alone in PTCL
Acronym: CRESCENDO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-Bel-301 Study; 70,789 (Other: FDA)
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — belinostat; 10-propargyl-10-deazaaminopterin; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Intervention Model Description: A Phase 3, Randomized, Open-Label Study Comparing the Efficacy and Safety of the Combination of Beleodaq-CHOP or Folotyn-COP to the CHOP Regimen Alone in Newly Diagnosed Patients with Peripheral T-Cell Lymphoma
Masking Description: None - Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1a (Active Comparator): Group 1a Belinostat 600 mg/m2 + CHOP
  Interventions: Drug: Belinostat Injection; Drug: CHOP
- Group 1b (Active Comparator): Group 1b Belinostat 1000 mg/m2 + CHOP
  Interventions: Drug: Belinostat Injection; Drug: CHOP
- Group 2a (Active Comparator): Group 2a Pralatrexate 20 mg/m2 + COP
  Interventions: Drug: Pralatrexate Injection; Drug: COP
- Group 2b (Active Comparator): Group 2b Pralatrexate 30 mg/m2 + COP
  Interventions: Drug: Pralatrexate Injection; Drug: COP
- Group 3 (Active Comparator): CHOP
  Interventions: Drug: CHOP

INTERVENTIONS:
Drug: Belinostat Injection — Belinostat 600 mg/m2 or 1000 mg/m2 along with CHOP is given in each cycle
  Other Names: Beleodaq®
  Arms: Group 1a; Group 1b
Drug: Pralatrexate Injection — Pralatrexate 20 mg/m2 or 30 mg/m2 along with COP is given in each cycle
  Other Names: Folotyn®
  Arms: Group 2a; Group 2b
Drug: CHOP — CHOP is the comparator arm
  Other Names: Cyclophosphamide, Hydroxydaunorubicin (doxorubicin), Oncovin (vincristine), and Prednisone
  Arms: Group 1a; Group 1b; Group 3
Drug: COP — COP is given in combination with Pralatrexate
  Other Names: Cyclophosphamide, Oncovin (vincristine), and Prednisone
  Arms: Group 2a; Group 2b

SUMMARY:
Part 1: This is a 5 Arm study primarily to determine the best dose out of the two dose levels of Belinostat and Pralatrexate combined with CHOP/COP in newly diagnosed PTCL patients based on Safety for part 2 study.

Part 2 (Efficacy and Safety): This is a 3 Arm study. Patients with previously untreated PTCL will be randomized 1:1:1 into 1 of 3 treatment groups: 2 experimental treatment groups (Bel-CHOP or Fol-COP) or 1 active comparator treatment group (CHOP). Patients will be treated for up to 6 cycles. The primary objective is to compare the Progression Free Survival of patients with newly diagnosed PTCL treated for up to 6 cycles with Beleodaq (belinostat) in combination with CHOP (Bel-CHOP) or Folotyn (pralatrexate injection) in combination with COP (Fol-COP) to CHOP alone.

DETAILED DESCRIPTION:
Study Design and Treatment Plan:

Part 1: Dose Finding

It is a randomized, open label, multicenter study in patients with PTCL who have not been previously treated and the control arm is CHOP, COP, is the CHOP regimen without Doxorubicin (H). Two investigational agents are separately added to C(H)OP, Belinostat for Bel-CHOP and Pralatrexate for FOL-COP. In this first part, each investigational arm will have two dose levels which will be compared with CHOP as reference. Treatment will be randomized in five arms:

1. Group 1a (Bel-CHOP) Belinostat 600 mg/m2
2. Group 1b (Bel-CHOP) Belinostat 1000 mg/m2
3. Group 2a (Fol-COP) Pralatrexate 20 mg/m2
4. Group 2b (Fol-COP) Pralatrexate 30 mg/m2
5. Group 3 for CHOP alone. Analysis will be done when 75 patients have received their planned treatment cycles to evaluate treatment compliance.

Approximately 20 patients will be enrolled into each group and receive at least one cycle of drug thus 15 patients are expected to be evaluated with their planned treatment of 6 cycles completed. The safety data will be evaluated to select the proper dose for Belinostat -CHOP and Pralatrexate-COP for the Part 2 study.

Part 2: Efficacy and Safety

It is a randomized, open-label, multicenter study in newly diagnosed PTCL patients. This is a three arm study and 143 patients will enroll in each arm. Patients will be randomized in a balance manner (1:1:1) into 1 of 3 treatment groups and treated for up to 6 cycles:

Group 1: (Bel-CHOP): Belinostat at the dose determined from Part 1 (600 or 1000 mg/m2) to be administered on Day 1 by 30 min intravenous (IV) infusion once daily for 5 days; CHOP will also be administered starting on Day 1 within 15 min (±5 min) after the end of the belinostat infusion at the doses shown below for Group 3, with cycles repeated every 21 days for up to 6 cycles

Group 2: (Fol-COP): Pralatrexate at the dose determined from part 1 (20 or 30 mg/m2) is to be administered on Day 1 and Day 8 as an IV push over 3 to 5 min; CHOP will also be administered starting on Day 1 within 15 min (±5 min) after the end of the pralatrexate administration at the doses shown below for Group 3, with cycles repeated every 21 days for up to 6 cycles. COP combination refers to CHOP without Doxorubicin (H).

Group 3: (CHOP): Combination chemotherapy to be administered starting on Day 1 at the doses shown below, with cycles repeated every 21 days for up to 6 cycles

* Cyclophosphamide 750 mg/m2 IV, Day 1
* Doxorubicin 50 mg/m2 IV, Day 1 (limit lifetime cumulative dose to <550 mg/m² to reduce risk of cardiotoxicity)
* Vincristine 1.4 mg/m2 (maximum 2 mg) IV, Day 1
* Prednisone 100 mg orally (PO) daily, Day 1 (after the end of the belinostat or pralatrexate administration for Groups 1 and 2) to Day 5

Randomization will be stratified on:

* Histology (nodal, extra-nodal)
* Prognostic Index for T-Cell Lymphoma (Group 1 or 2 vs 3 or 4)
* Region (US, ex-US)

The study duration will include up to a 28-day screening period, a 6-cycle treatment period (18 weeks), follow-up until progression, an End-of-Treatment Visit at least 30 days after the last dose of study treatment, and long-term survival follow-up for patients by phone every 6 months thereafter until a 5-year median follow-up of the population is reached. Patients discontinuing the study for other reasons than progression will have the same long-term follow-up for OS analysis. Tumor assessments will be performed every 3 cycles (i.e., 9 weeks) on Cycle 4 Day 1 and End-of-Treatment Visit during treatment, then every 3 months for 3 years for patients with complete response (CR), partial response (PR), or stable disease, and every 6 months thereafter until disease progression or death

ELIGIBILITY:
Inclusion Criteria:

1. Patient with newly diagnosed, untreated histology-proven PTCL based on local pathology review who is eligible for receiving, Belinostat, Pralatrexate, and CHOP. Pathology material must be available at the site for each patient before enrollment so that it can be sent to the Sponsor (or designee) for later confirmation. The following subtypes, as defined by the updated World Health Organization (WHO) classification, may be included. This information should be available for eligibility:

   1. Pathology subtype:

      * Peripheral T-cell lymphoma, not otherwise specified
      * Angioimmunoblastic T-cell lymphoma
      * Anaplastic lymphoma kinase (ALK)-negative anaplastic large-cell lymphoma (ALCL) patients are eligible only if Brentuximab Vedotin (BV) is not commercially approved for use, not available in the country or patient is contraindicated to receive BV.
      * Follicular T-cell lymphoma
      * Others: Extra-nodal natural killer/T-cell lymphoma, nasal type; enteropathy-associated T-cell lymphoma; hepatosplenic T-cell lymphoma; and subcutaneous panniculitis-like T-cell lymphoma
   2. CD30 expression and T-cell Follicular Helper (TFH) phenotype status must be available for documentation.
2. Patient has at least 1 site of measurable disease according to Response Evaluation Criteria in Lymphoma (RECIL) 2017 criteria as assessed by the local Investigator (Appendix 3)
3. Patient has an Eastern Cooperative Oncology Group performance (ECOG) status ≤2
4. For Part 1 (Dose Finding) - Patient has adequate hematological, hepatic, and renal function as defined by:

   1. Absolute neutrophil count ≥ 1.5 × 10⁹/L or ≥ 1.0 × 10⁹/L if evidence of bone marrow involvement
   2. Platelet count ≥100×10⁹/L or ≥ 75×10⁹/L if evidence of bone marrow involvement
   3. Total bilirubin ≤1.5 mg/dL
   4. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 3×upper limit of normal (ULN; AST/ALT ≤5×ULN if documented hepatic involvement with lymphoma)
   5. Calculated creatinine clearance of ≥ 60 mL/min
5. Part 2 (Efficacy and Safety) - disease related hypoplasia, hepatological or renal dysfunction can be included if any of the treatment groups can be administered based on package insert recommendation with the following restrictions:

   1. Absolute neutrophil count ≥ 1.5 × 10⁹/L or ≥ 1.0 × 10⁹/L if evidence of bone marrow involvement
   2. Platelet count ≥100×10⁹/L or ≥ 75×10⁹/L if evidence of bone marrow involvement
   3. Total bilirubin ≤1.5 mg/dL
   4. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤ 3 x the upper limit of normal (ULN; AST/ALT ≤5×ULN if documented hepatic involvement with lymphoma)
   5. Calculated creatinine clearance of ≥ 60 mL/min
6. UGT1A1 genotype has been characterized (see Belinostat dose modifications if abnormal) and must be available for documentation.
7. Patient must be willing and capable of giving written informed consent and must be able to adhere to dosing and visit schedules and meet all study requirements
8. Patient (male or female) is at least 18 years of age at the time of informed consent
9. Patient is willing to practice 2 forms of contraception, one of which must be a barrier method, from study entry until at least 6 months after the last dose of study treatment.
10. Females of childbearing potential must have a negative urine pregnancy test within 4 weeks prior to the first day of study treatment. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or are surgically sterilized do not require this test.

Exclusion Criteria:

A patient will not be eligible for inclusion if ANY of the criteria listed below apply:

1. Patients with a diagnosis of:

   1. Precursor T-cell lymphoma or leukemia
   2. Adult T-cell lymphoma/leukemia
   3. T-cell prolymphocytic leukemia
   4. T-cell large granular lymphocytic leukemia
   5. Primary cutaneous type ALCL
   6. Cutaneous T-cell lymphoma (mycosis fungoides/Sezary syndrome)
   7. ALCL if they can be treated with Brentuximab Vedotin (BV)
2. Patients taking drugs which are potent UGT1A1 inhibitors must discontinue one week before randomization; drug can be resumed if the treatment doesn't include belinostat
3. Patient with an active concurrent malignancy/life-threatening disease with the exception of non melanoma skin tumors and in situ cervical cancer if they have received treatment resulting in complete resolution of the cancer and currently have no clinical, radiologic, or laboratory evidence of active or recurrent disease. If there is a history of prior malignancies/life-threatening diseases, the patient must be disease free for at least 5 years
4. Prior histone deacetylase (HDAC) inhibitor or pralatrexate therapy
5. Any known cardiac abnormalities such as baseline prolongation of QT/corrected QT (QTc) interval (i.e. demonstration of a QTc interval >450 msec); long QT syndrome; myocardial infarction within 6 months prior to starting study; history of significant cardiovascular disease; the required use of a concomitant medication that may cause Torsades de Pointes
6. Patient with uncontrolled hypertension
7. Patients status on the following:

   1. Has a known HIV-positive diagnosis with uncontrolled and detectable viral load
   2. Has Hepatitis B or Hepatitis C virus diagnosis with uncontrolled and detectable viral load or immunological evidence of chronic active disease
8. Patient with central nervous system metastasis
9. Patient with an active uncontrolled infection, underlying medical condition, laboratory abnormality, or other serious illness that would impair the ability of the patient to receive protocol treatment
10. Patient who has used any investigational drugs, biologics, or devices within 28 days prior to study treatment or plans to use any of these during the course of the study
11. Patient with a known history of drug or alcohol abuse
12. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
PFS | 4.5 years
  Progression-free survival is determined from randomization to the first documented Progression of Disease or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 8 years
  It is the time from randomization to the death

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srinivas Atmuri, MPharm, MS, Study Director — Acrotech Biopharma Inc.
Locations (69):
- United States (11):
  - University of California, San Francisco Fresno, Clovis, California
  - University of California, Los Angeles Hem/ Onc Clinical Research Unit, Suite 600, Santa Monica, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Moffitt Malignant Hematology & Cellular Therapy at Memorial Healthcare System Memorial Cancer Institute, Pembroke Pines, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Valley Cancer Associates, Harlingen, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Germany (2):
  - Universitatsmedizin Gottingen, Göttingen
  - Universitaetsklinikum Halle (Saale), Halle
- Hungary (6):
  - University of Debrecen Clinical Center, Debrecen, Nagyerdei Krt. 98
  - Andras Josa University Teaching Hospital, Nyíregyháza, Szent Istvan Utca
  - Semmelweis Egyetem, Budapest
  - National Institute of Oncology, Budapest
  - Markhot Ferenc Oktato Korhaz, Eger
  - Belgyogyaszati Klinika es Kardiologiai Kozpont, Szeged
- Italy (9):
  - Azienda Ospedaliera Cardinale Giovanni Panico, Tricase, Apulia
  - University of Milano Bicocca, Milan, Bicocca
  - Servizio Sanitario Regionale Emilia-Romagna-Istituto Scientifico Romagnolo per lo Studio dei Tumori "Dino Amadori" Srl (IRST), Meldola, Province Of Forlì-Cesena
  - Policlinico GB Rossi Borgo Roma, Borgo Roma, Verona
  - Azienda Ospedaliera SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Ospedale Policlinico San Martino, IRCCS, Genova
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda USL di Ravenna, Ravenna
- Poland (4):
  - University Hospital in Wroclaw, Wroclaw, Wroclaw
  - Pratia MCM Krakow, Krakow
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship
- South Korea (13):
  - Inje University Busan Paik Hospital, Busan, Busanjin District
  - Ulsan University Hospital, Ulsan, Dong-gu
  - Ajou University Hospital, Suwon, Gyenoggi-do
  - The Catholic University of Korea - St. Vincents Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Yeungnam University Medical Center, Daegu, Nam-gu
  - Severance hospital, Yonsei University, Sinchon-dong, Seoul
  - Asan Medical Center, Songpa-dong, Seoul
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (10):
  - Hospital Universitario Basurto, Bilbao, Bizkaia
  - Hospital Universitario Fundación Jiménez Díaz, Moncloa-Aravaca, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital del Mar Medical Research Institute, Barcelona
  - ICO - Hospital Duran i Reynals, Barcelona
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - Changhua Christian Hospital CCH, Changhua, Changhua County
  - Hualien Tzu Chi Medical Center, Hualien City, Hualien
  - National Cheng Kung University Hospital NCKUH, Tainan, Southern Taiwan
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - Hematology Oncology Taipei Medical University - Shuang-Ho Hospital, New Taipei City
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Turkey (Türkiye) (6):
  - Ankara University Medical Faculty Hospital, Altındağ, Ankara
  - Bilkent University, Çankaya, Ankara
  - Gazi University Faculty of Medicine, Yenimahalle, Ankara
  - VKV AMERICAN HOSPITAL, Medical Oncology Outpatient Clinic, Şişli, Istanbul
  - Adana City Education and Research Hospital, Adana
  - Ege Univ. Hospital, Bornova

IPD SHARING:
Plan to Share IPD: No
Data Review Committee:
  An Independent Data Monitoring Committee (IDMC) will be established for the purpose of reviewing patient safety and the results of the futility analysis. The IDMC will convene after the enrollment and analysis of Part 1 to evaluate safety and preliminary efficacy. The IDMC will recommend the selected dose for Belinostat and Pralatrexate. The IDMC will also convene after the analysis of 120 events, in Part 2, to state whether the study can continue.
  This Committee will review review study data will adjudicate tumor response and the date of onset of disease progression in all patients at the end of the study. All scans will be centrally reviewed and the primary analysis of PFS will be conducted on these results.